CLINICAL TRIAL: NCT04296396
Title: Prescription After Cesarean Trial
Brief Title: Opioid Prescription After Cesarean Trial
Acronym: PACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HD036801-PACT; U24HD036801 (NIH); UG1HD087230 (NIH); UG1HD027869 (NIH); UG1HD027915 (NIH); UG1HD034208 (NIH); UG1HD040500 (NIH); UG1HD040485 (NIH); UG1HD053097 (NIH); UG1HD040544 (NIH); UG1HD040545 (NIH); UG1HD040560 (NIH); UG1HD040512 (NIH); UG1HD087192 (NIH)
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Pregnancy Related; Opioid Use; Pain
MeSH Terms: conditions — Pain | interventions — Oxycodone

STUDY DESIGN:
Intervention Model Description: Participants were randomized to either an individualized opioid prescription protocol (IOPP) that includes shared decision making or to a fixed opioid prescription of 20 tablets of oxycodone 5mg.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Individualized Opioid Prescription (Experimental): Individualized opioid prescription protocol and shared decision making
  Interventions: Drug: 0 to 20 tablets of oxycodone 5mg
- Fixed Opioid Prescription (Other): Fixed opioid prescription of 20 tablets of oxycodone 5mg
  Interventions: Drug: Fixed opioid prescription

INTERVENTIONS:
Drug: 0 to 20 tablets of oxycodone 5mg — Individualized opioid prescription protocol (IOPP) that includes shared decision making
  Arms: Individualized Opioid Prescription
Drug: Fixed opioid prescription — 20 tablets of oxycodone 5mg
  Arms: Fixed Opioid Prescription

SUMMARY:
Non-inferiority randomized trial of 5,500 women with a cesarean delivery randomized prior to discharge to either an individualized opioid prescription protocol (IOPP) that includes shared decision making or to a fixed opioid prescription of 20 tablets of oxycodone 5mg.

DETAILED DESCRIPTION:
This was a non-inferiority multi-center unblinded randomized trial of 5,500 women undergoing a cesarean delivery who were randomized before discharge to either an individualized opioid prescription protocol (IOPP) that includes shared decision making or to a fixed opioid prescription of 20 tablets of oxycodone 5mg. The primary endpoint was the presence/absence of moderate to severe pain at 1 week after discharge. Moderate to severe pain was defined as a value of 4 or higher on the Brief Pain Inventory worst pain scale (0 to 10) in the last 24 hours. Consenting women were assigned in a 1:1 ratio to one of the two arms using a secure internet based randomization system maintained centrally by the Data Coordinating Center (DCC). Randomization was stratified by site. Women were followed through 90 days postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Post cesarean delivery (combined vaginal/cesarean deliveries are not eligible)
* Singleton, twin or triplet gestation

Exclusion Criteria:

* An opioid prescription filled during the current pregnancy
* Known history of opioid use disorder, by medical record review
* Contraindication to opioids (oxycodone)
* Contraindications to both acetaminophen and ibuprofen
* Significant surgical procedures (e.g., hysterectomy) prior to randomization as pain trajectory will be completely different
* Fetal or neonatal death prior to randomization
* Inability to randomize within 1 day before planned discharge from the hospital
* Inability to participate in shared decision making as assessed by research staff
* Language barrier (non-English or Spanish speaking)
* Participation in this trial in a previous pregnancy
* Participation in another intervention study that influences the primary outcome in this trial

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5521 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Longo, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (12):
- United States (12):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Columbia University, New York, New York
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve-Metrohealth, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Brown Univeristy, Providence, Rhode Island
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be shared per NIH policy after the completion and publication of the main analyses. Data will be available through the NICHD Data and Specimen Hub.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Smid MC, Clifton RG, Rood K, Srinivas S, Simhan HN, Casey BM, Longo M, Landau R, MacPherson C, Bartholomew A, Sowles A, Reddy UM, Rouse DJ, Bailit JL, Thorp JM Jr, Chauhan SP, Saade GR, Grobman WA, Macones GA; for the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network*. Optimizing Opioid Prescription Quantity After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2024 Aug 1;144(2):195-205. doi: 10.1097/AOG.0000000000005649. Epub 2024 Jun 10. PMID 38857509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We conducted this multicenter, randomized, controlled, double blinded trial at 31 hospitals. From September 2020 through March 2022, a total of 18,990 patients underwent screening for randomization. Of the 9,963 eligible patients, 5,521 provided informed consent and were randomized
Pre-assignment Details: 1 participant in the Fixed Opioid Prescription Arm/Group was reenrolled in the study for a second pregnancy
Groups:
- Individualized Opioid Prescription Protocol (IOPP): Individualized opioid prescription protocol (IOPP) with shared decision making. IOPP will be based on inpatient oral opioid intake during the 24 hour period prior to randomization and should not include the 12 hours immediately after the cesarean.
- Fixed Opioid Prescription: Fixed amount of opioids (20 tablets of oxycodone 5mg)
Period: Overall Study
Arm/Group | Individualized Opioid Prescription Protocol (IOPP) | Fixed Opioid Prescription
Started | 2748 | 2773
Completed (Participants who completed the 90 day visit.) | 2386 | 2426
Not Completed | 362 | 347

BASELINE CHARACTERISTICS:
Population: Baseline data were collected once for the one participant who re-enrolled
Groups:
- Individualized Opioid Prescription: Individualized opioid prescription protocol (IOPP) with shared decision making
  IOPP will be based on inpatient oral opioid intake during the 24 hour period prior to randomization and should not include the 12 hours immediately after the cesarean.
- Total: Total of all reporting groups
Arm/Group | Individualized Opioid Prescription | Fixed Opioid Prescription | Total
Number analyzed (Participants) | 2748 | 2772 | 5520
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data is missing for one participant in each group.
  years
    number analyzed (Participants) | 2747 | 2771 | 5518
    (all) | 30.5 (5.7) | 30.3 (5.8) | 30.4 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2748 | 2772 | 5520
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity Customized: American Indian/Alaskan Native | 24 | 17 | 41
  Race/Ethnicity Customized: Asian | 118 | 119 | 237
  Race/Ethnicity Customized: Non-Hispanic Black | 759 | 746 | 1505
  Race/Ethnicity Customized: Hispanic | 574 | 589 | 1163
  Race/Ethnicity Customized: Native Hawaiian/Pacific Islander | 9 | 7 | 16
  Race/Ethnicity Customized: Non-Hispanic White | 1158 | 1194 | 2352
  Race/Ethnicity Customized: More than one race | 72 | 78 | 150
  Race/Ethnicity Customized: Unknown/Not Reported | 34 | 22 | 56
Number of cesarean deliveries [Count of Participants; unit: Participants] — The number of cesarean deliveries, including the birth during this hospital admission. Population: Data is missing for one participant from each group.
  Participants
    number analyzed (Participants) | 2747 | 2771 | 5518
    One | 1623 | 1630 | 3253
    Two | 730 | 735 | 1465
    Three or more | 394 | 406 | 800
Type of labor [Count of Participants; unit: Participants] — The type of labor experienced for the birth during the current hospital admission. Population: Data is missing for one participant in each group.
  Participants
    number analyzed (Participants) | 2747 | 2771 | 5518
    No labor | 1411 | 1392 | 2803
    Spontaneous | 558 | 574 | 1132
    Induced | 778 | 805 | 1583

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Worst Pain Score of Moderate to Severe on the Brief Pain Inventory
Description: Number of participants with moderate to severe pain at 1 week post-discharge; moderate to severe pain is defined as a value of 4 or higher on the "Worst Pain" question of the Brief Pain Inventory (BPI) in the last 24 hours. The BPI measures pain severity on a numeric scale of 0 to 10, with 0 being no pain and 10 being the highest level of pain.
Time Frame: 1 week post hospital discharge
Population: Of 2273 participants in the fixed group, 1 was enrolled in the study for a second pregnancy. Only the first pregnancy was included in the analysis. The primary analysis included participants who completed the highest pain in the last 24 hours on the Brief Pain Inventory at 1 week post-discharge. This data was missing for 230 participants in the individualized opioid prescription group and 219 participants in the fixed group.
Measure: Count of Participants; unit: Participants
Groups:
- Individualized Opioid Prescription: Individualized opioid prescription protocol and shared decision making
  0 to 20 tablets of oxycodone 5mg: Individualized opioid prescription protocol (IOPP) that includes shared decision making. IOPP will be based on inpatient oral opioid intake during the 24 hour period prior to randomization and should not include the 12 hours immediately after the cesarean.
Arm/Group | Individualized Opioid Prescription | Fixed Opioid Prescription
Number analyzed (Participants) | 2518 | 2553
Participants | 1497 | 1535
Statistical Analysis 1: Comparison: Individualized Opioid Prescription vs Fixed Opioid Prescription; Test type: Non-Inferiority — A non-inferiority design assumed a noninferiority margin of 5%. For 90% power and 0.025 significance level 1-sided, a total sample size of 4,300 participants was required to state that the IOPP is not inferior to the fixed amount of 20 tablets. Given the short window to assess pain at 1-week post-discharge, a 20% missing rate was incorporated which gives a final sample size of 5,500 (2,750 per group); Risk Difference (RD) = 0.67, 95% CI 2-sided [-2.03 to 3.37] — The risk difference is the rate in the fixed group minus the rate in the IOPP group. IOPP was to be determined as non-inferior if the lower 95% confidence limit for the risk difference is -5 percentage points or greater (i.e., closer to zero)

2. Secondary Outcome: Number of Participants Who Filled One or More Opioid Prescriptions Beyond the Amount Prescribed at Discharge
Description: Number of participants who filled one or more opioid prescriptions beyond what was prescribed to them at discharge - measured at ninety days postpartum
Time Frame: After hospital discharge and up to 90 days postpartum
Population: Of 2273 participants in the fixed group, 1 was enrolled in the study for a second pregnancy. Only the first pregnancy was included in the analysis. This data was missing for 94 participants in the individualized opioid prescription group and 76 participants in the fixed group.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Opioid Prescription | Fixed Opioid Prescription
Number analyzed (Participants) | 2654 | 2696
Participants | 200 | 166
Statistical Analysis 1: Comparison: Individualized Opioid Prescription vs Fixed Opioid Prescription; Test type: Superiority; p = 0.046, Chi-squared; Risk Ratio (RR) = 1.22, 96.25% CI 2-sided [0.99 to 1.51] — Confidence interval is 96.25% due to false discovery rate adjustment

3. Secondary Outcome: Number of Opioid Prescriptions Filled
Description: Number of opioid prescriptions filled by ninety days postpartum
Time Frame: 90 days postpartum
Population: 94 missing in the IOPP group. 75 missing in the fixed group
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Opioid Prescription Protocol (IOPP) | Fixed Opioid Prescription
Number analyzed (Participants) | 2654 | 2697
Participants
  Number of participants who filled zero prescriptions | 601 | 452
  Number of participants who filled one prescription | 1873 | 2086
  Number of participants who filled 2 prescriptions | 163 | 140
  Number of participants who filled 3 prescriptions | 12 | 16
  Number of participants who filled 4 prescriptions | 5 | 3
Statistical Analysis 1: Comparison: Individualized Opioid Prescription Protocol (IOPP) vs Fixed Opioid Prescription; Test type: Superiority; p < 0.001, Chi-squared

4. Secondary Outcome: Number of Opioid Tablets Unused Since Discharge
Description: Number of opioid tablets unused from discharge to 90 days postpartum
Time Frame: 90 days postpartum
Population: Data were missing for 207 participants in the IOPP group and for 180 in the fixed group.
Measure: Median (Inter-Quartile Range); unit: tablets
Arm/Group | Individualized Opioid Prescription | Fixed Opioid Prescription
Number analyzed (Participants) | 2541 | 2592
tablets | 2 [0 to 8] | 7 [0 to 16]
Statistical Analysis 1: Comparison: Individualized Opioid Prescription vs Fixed Opioid Prescription; Test type: Superiority; p < 0.001, quantile regression; Median Difference (Net) = -5, 97.5% CI 2-sided [-6.6 to -3.5] — Confidence interval is 97.5% due to false discovery rate adjustment

5. Secondary Outcome: Number of Morphine Milligram Equivalents Used at 2 Weeks Post Discharge
Description: Total morphine milligram equivalents (MME) used from discharge to 2 weeks post-discharge. MME is the amount of milligrams of morphine an opioid dose is equal to when prescribed. Calculating MME accounts for differences in opioid drug type and strength.
Time Frame: 2 weeks post discharge
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalent
Arm/Group | Individualized Opioid Prescription | Fixed Opioid Prescription
Number analyzed (Participants) | 2748 | 2772
morphine milligram equivalent | 22.5 [0 to 75.0] | 37.5 [0 to 97.5]
Statistical Analysis 1: Comparison: Individualized Opioid Prescription vs Fixed Opioid Prescription; Test type: Superiority; p < 0.001, quartile regression; Median Difference (Net) = -15, 98.75% CI 2-sided [-19.2 to -10.8] — Confidence interval is 98.75% due to false discovery rate adjustment

6. Secondary Outcome: Worst Pain Severity Score at 2 Weeks Post Discharge
Description: Pain severity scores assessed on the Brief Pain Inventory numeric scale from 0 to 10 at 2 weeks post-discharge. The BPI measures pain severity on a numeric scale of 0 to 10, with 0 being no pain and 10 being the highest level of pain.
Time Frame: 2 weeks post discharge
Population: Data were missing for 234 participants in the IOPP group and for 286 in the fixed group
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Individualized Opioid Prescription Protocol (IOPP) | Fixed Opioid Prescription
Number analyzed (Participants) | 2514 | 2486
score on a scale | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0]
Statistical Analysis 1: Comparison: Individualized Opioid Prescription Protocol (IOPP) vs Fixed Opioid Prescription; Test type: Superiority; p = 1.0, quantile regression; Median Difference (Net) = 0, 95% CI 2-sided [0 to 0]

7. Secondary Outcome: Pain Interference Score ≥ 4 at 2 Weeks Post Discharge
Description: Pain interference scores ≥ 4 on the Brief Pain Inventory (numeric scale from 0 to 10) at 2 weeks post-discharge. The BPI measures pain severity on a numeric scale of 0 to 10, with 0 being no pain and 10 being the highest level of pain. This outcome asks participants to indicate their pain scores for the week prior to completing the inventory.
Time Frame: 2 weeks post discharge
Population: Data were missing for 234 participants in the IOPP group and for 286 in the fixed group
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Opioid Prescription Protocol (IOPP) | Fixed Opioid Prescription
Number analyzed (Participants) | 2514 | 2486
Participants | 415 | 427
Statistical Analysis 1: Comparison: Individualized Opioid Prescription Protocol (IOPP) vs Fixed Opioid Prescription; Test type: Superiority; p = 0.52, Chi-squared; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.85 to 1.09]

8. Secondary Outcome: Number of Participants Who Indicated an Improved Global Impression of Change
Description: Number of participants who indicated an improved global impression of change in overall pain at 2 weeks post-discharge. This represents a selection on a multiple choice survey question with the response options: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse.
Time Frame: 2 weeks post discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Opioid Prescription Protocol (IOPP) | Fixed Opioid Prescription
Number analyzed (Participants) | 2528 | 2509
Participants | 2436 | 2436
Statistical Analysis 1: Comparison: Individualized Opioid Prescription Protocol (IOPP) vs Fixed Opioid Prescription; Test type: Superiority; p = 0.15, Regression, Linear; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.98 to 1.00]

9. Secondary Outcome: Infant Hospital Readmissions
Description: Proportion of infants readmitted to the hospital
Time Frame: 6 weeks postpartum
Population: 2856 and 2889. Data is missing for 102 neonates in the IOPP group and 92 neonates in the fixed opioid group.
Measure: Count of Participants; unit: Participants
Groups:
- Individualized Opioid Prescription (IOPP) -Neonates/Infants: Neonates/infants of participants in the Individualized opioid prescription protocol (IOPP) with shared decision making group.
- Fixed Opioid Prescription - Neonates/Infants: Neonates/infants of participants in the fixed opioid prescription group.
Arm/Group | Individualized Opioid Prescription (IOPP) -Neonates/Infants | Fixed Opioid Prescription - Neonates/Infants
Number analyzed (Participants) | 2754 | 2793
Participants | 59 | 63

10. Secondary Outcome: Maternal Depression Score ≥ 13
Description: The proportion of participants with a score of 13 or higher on the Edinburgh Postnatal Depression Scale. The minimum score is 0 and the maximum score is 30. Higher scores indicate worse outcomes, where persons scoring about 13 are likely to be suffering from a depressive illness. The scale indicates how the respondent has felt during the previous week.
Time Frame: 6 weeks postpartum
Population: data is missing for 252 participants in the IOPP group and 276 participants in the fixed prescription group
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Opioid Prescription Protocol (IOPP) | Fixed Opioid Prescription
Number analyzed (Participants) | 2496 | 2496
Participants | 185 | 191

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of randomization at delivery through 90 days postpartum (a period of 90 days). Adverse events were collected for maternal participants and their neonates.
Groups:
- Individualized Opioid Prescription (IOPP) -Mother: Individualized opioid prescription protocol (IOPP) with shared decision making. IOPP will be based on inpatient oral opioid intake during the 24 hour period prior to randomization and should not include the 12 hours immediately after the cesarean.
- Fixed Opioid Prescription -Mother: Fixed amount of opioids (20 tablets of oxycodone 5mg)
Arm/Group | Individualized Opioid Prescription (IOPP) -Mother | Fixed Opioid Prescription -Mother | Individualized Opioid Prescription (IOPP) -Neonates/Infants | Fixed Opioid Prescription - Neonates/Infants
All-Cause Mortality (participants affected / at risk) | 0/2748 | 0/2772 | 11/2856 | 8/2889
Serious Adverse Events (participants affected / at risk) | 133/2748 | 96/2772 | 37/2856 | 30/2889
Other Adverse Events (participants affected / at risk) | 166/2748 | 186/2772 | 0/2856 | 0/2889
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individualized Opioid Prescription (IOPP) -Mother (N=2748) | Fixed Opioid Prescription -Mother (N=2772) | Individualized Opioid Prescription (IOPP) -Neonates/Infants (N=2856) | Fixed Opioid Prescription - Neonates/Infants (N=2889)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — includes cardiac arrest and coarctation of aorta
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angiodysplasia of duodenum (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Neonatal death (General disorders) | 0 (0) | 0 (0) | 10 (10) | 8 (8)
Polydactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mastitis (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Abdominal adhesions (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heavy vaginal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal fluid collection (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postpartum endometritis (Reproductive system and breast disorders) | 8 (8) | 9 (9) | 0 (0) | 0 (0)
Septic pelvic thrombophlebitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Myocardial infarction type 2 (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
New onset diastolic heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraparenchymal hemorrhage (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lower extremity swelling (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous thromboembolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystectomy (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Distal bowel stricture (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intrauterine bowel perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meconium pseudocyst and volvulous (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Poor feeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Poor weight gain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pale/Stiff (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suspected congenital adrenal hyperplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trisomy 18 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coarctation of aorta (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (6) | 6 (7)
Hypospadias (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalomalacia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Seizures (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Glioblastoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postpartum preeclampsia (Pregnancy, puerperium and perinatal conditions) | 62 (63) | 54 (56) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (5) | 3 (3)
Escherichia coli cystitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5) | 0 (0) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incisional bleeding (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Skin and subcutaneous tissue disorders) | 23 (25) | 10 (11) | 0 (0) | 0 (0)
Hypothermia (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Choledocholithiasis (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individualized Opioid Prescription (IOPP) -Mother (N=2748) | Fixed Opioid Prescription -Mother (N=2772) | Individualized Opioid Prescription (IOPP) -Neonates/Infants (N=2856) | Fixed Opioid Prescription - Neonates/Infants (N=2889)
Drowsiness (General disorders) | 166 (166) | 186 (186) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT04296396/Prot_SAP_001.pdf